CLINICAL TRIAL: NCT06490094
Title: Impact of Inquiry-Based Stress Reduction (IBSR) on Postpartum Mothers' Mental Health.
Brief Title: Impact of IBSR on Postpartum Mothers' Mental Health.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, shahar lev-ari, Impact of Inquiry-Based Stress Reduction (IBSR) on Postpartum Mothers' Mental Health., Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBSR Postpartum Mothers
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Postpartum Mothers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inquiry Based Stress Reduction (Experimental): Inquiry Based Stress Reduction (IBSR) program
  Interventions: Behavioral: Inquiry Based Stress Reduction (IBSR)
- Control group (No Intervention): Postpartum mothers who are randomly assigned to not receive the Inquiry-Based Stress Reduction (IBSR) intervention

INTERVENTIONS:
Behavioral: Inquiry Based Stress Reduction (IBSR) — The 8-week IBSR program is a clinical intervention based on "The Work" method, developed by Byron Katie and run in the US and Europe for 35 years. The IBSR intervention will involve weekly group meetings (3 hours/meeting) throughout 8 weeks. Home practice between sessions will be supported by facilitator assistants (1-hour session per week). All sessions will be standardized according to the IBSR certification program guidelines and will be assessed to maintain consistency in the program, as in previous studies. .
  Arms: Inquiry Based Stress Reduction

SUMMARY:
The period of pregnancy, childbirth, and the postpartum phase significantly impacts the mental health of women and their families. Mental health is crucial for overall well-being, quality of life, and is associated with healthcare costs. Therefore, promoting mental health should be a top priority in public health and health promotion efforts.

The Inquiry-Based Stress Reduction (IBSR) intervention, developed by Byron Katie ("The Work"), enables participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR involves a contemplative "inquiry" process and a "turnaround," which is a method of experiencing the opposite of what the participant believes. This process equips individuals with skills for self-inquiry and management of stressful thoughts that can be easily integrated into daily life.

Based on previous research, we hypothesize that the IBSR intervention can improve postpartum mothers' mental health.

DETAILED DESCRIPTION:
In recent years, there is growing evidence regarding the effectiveness of population-based mental health promotion interventions. Developing social and emotional skills such as improved self-esteem, sense of control and self-efficacy, self-acceptance, purpose in life, positive relationships with others, problem-solving, and coping skills has been shown to improve mental health and contribute to psychological well-being. According to the International Union for Health Promotion and Education (IUHPE, 2021), interventions to promote mental health can be classified into eight priority areas. The first priority is to promote the mental health of infants and mothers by focusing on social and emotional development and positive mental health in early childhood development services, including prenatal care, home visits, and parenting programs. The healthcare system today faces the challenge of gaining a better understanding of the mechanisms that allow women to develop and maintain positive mental health in the postpartum period and understanding how these mechanisms are sustained over time.

The Inquiry-Based Stress Reduction (IBSR) intervention, developed by Byron Katie ("The Work"), enables participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR involves a contemplative "inquiry" process and a "turnaround," which is a method of experiencing the opposite of what the participant believes. This process equips individuals with skills for self-inquiry and management of stressful thoughts that can be easily integrated into daily life. Based on previous research, we hypothesize that the IBSR intervention can improve postpartum mothers' mental health.

ELIGIBILITY:
Inclusion Criteria:

* Mothers up to two years after giving birth, between the ages of 18 and 45 (at the time of birth), without a history of mental disorders or illnesses

Exclusion Criteria:

* Mothers with a history of illness or mental disorders
* mothers who have passed more than two years since their last birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — postpartum mothers
Enrollment: 68 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Connor-Davidson Resilience Scale (2-item CD-RISC) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Ryff scale- Psychological well-being (PWB) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Subjective well-being (WHO-5) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Multidimensional Scale of Perceived Social Support (MSPSS) | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire

OTHER OUTCOMES:
Primary Care PTSD DSM-5 | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
exposure to the events of the war in Israel | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire
Demographic and Childhood history | A measure assessing change between 3 time points (before the intervention, after 2 months (at the end of the intervention) and 1 months later)
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lev- Ari, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No